CLINICAL TRIAL: NCT02005588
Title: Comparison Between Aminoacid Chelated Iron and Iron Salt in Treatment of Iron Deficiency Anemia With Pregnancy
Brief Title: Treatment of Iron Deficiency Anemia With Pregnancy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Abdel Fattah, lecturer of obstetrics and gynecology, faculty of medicine, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ferrot2013; nerhado pharmaceutical company (Registry Identifier: nerhado pharmaceutical company)
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: amino acid chelated iron; iron salt; iron deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- amino acid chelated iron arm (Active Comparator): this arm will contain 150 pregnant women with proved iron deficiency anemia and pregnant 14-18 weeks. these pregnant women will be given amino acid chelated iron capsules (15 mg iron/capsule) 1-2 capsules daily according to hemoglobin level (hemoglobin 7-9 g/dl will receive 2 capsules, and hemoglobin 9.1-11 g/dl will receive 1 capsule). complete blood picture and serum ferritin will be assessed at 22-23 weeks, 29-30 weeks and 36-37 weeks. possible side effects (colicky abdominal pains, constipation and metallic taste) will be asked about in each follow up visit.
  Interventions: Drug: amino acid chelated iron; Drug: iron salt (ferrous fumarate)
- iron salt arm (Active Comparator): this arm will contain 150 pregnant women with proved iron deficiency anemia and 14-18 weeks gestation. these women will be given oral iron salt ferrous fumarate capsules (350 mg iron/ capsule containing about 70 mg elemental iron/ capsule) 1-2 capsules daily according to hemoglobin level (hemoglobin 7-9 g/dl will receive 2 capsules daily and hemoglobin 9.1-11 g/dl will receive 1 capsule daily. women will be followed up with complete blood picture and serum ferritin at 22-23 weeks, 29-30 weeks and 36-37 weeks. women will be asked about possible side effects (colicky abdominal pains, constipation, and metallic taste) in each visit.
  Interventions: Drug: amino acid chelated iron; Drug: iron salt (ferrous fumarate)

INTERVENTIONS:
Drug: amino acid chelated iron — the drug will be given to pregnant women 14-18 weeks' gestation who prove to have iron deficiency anemia. the dose will be given according to hemoglobin level. for hemoglobin 7-9 g/dl, 2 capsules will be given daily. for hemoglobin 9.1-11 g/dl, 1 capsule will be given daily. complete blood picture and serum ferritin will be measured at 22-23, 29-30 and 36-37 weeks' gestation.
  Other Names: ferrotron capsules
Drug: iron salt (ferrous fumarate) — this drug will be given to pregnant women 14-18 weeks' gestation with iron deficiency anemia. the dose will be given according to hemoglobin level. for hemoglobin 7-9 g/dl, 2 capsules will be given daily, and for hemoglobin 9.1-11 g/dl, 1 capsule will be given daily. complete blood picture and serum ferritin will be measured at 22-23, 29-30 and 36-37 weeks' gestation.
  Other Names: hemoton capsules

SUMMARY:
Iron deficiency anemia is a very common problem accompanying pregnancy. in this study, the investigators are going to compare the efficacy and tolerability of two preparations of oral iron in treatment of iron deficiency anemia with pregnancy.

DETAILED DESCRIPTION:
In this study, the investigators are going to compare two preparations of oral iron in treatment of iron deficiency anemia with pregnancy. a total of 300 pregnant women will be randomly divided into two equal groups (each containing 150 pregnant woman). one group will receive amino acid chelated iron and the other group will receive iron salt (ferrous fumarate). All pregnant women attending the obstetrics outpatient clinic of kasr al aini hospital at 14-18 weeks gestation will be submitted to complete blood picture and serum ferritin. those who prove to have iron deficiency anemia (hemoglobin less than 11g/dl and serum ferritin less than 12ug/l) will be included in the study. All eligible women will be followed up at 22-23, 29-30 and 36-37 weeks' gestation for the change in hemoglobin level and ferritin level. all women will be also enquired about different side effects during treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years
* Pregnant 14-18 weeks
* Singleton fetus
* Hb 7-10.9 g/dl
* Serum ferritin <12 microgram/L

Exclusion Criteria:

* history of anemia due to other causes as chronic blood loss, hemolytic anemia or thalassemia
* Multiple pregnancy
* known hepatic, renal or cardiovascular abnormality.
* Known peptic ulcer, esophagitis, gastritis or hiatus hernia.
* Family history of thalassemia, sickle cell anemia, or malabsorption syndrome.
* Iron preparation intake within 24 hours of inclusion

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
change in hemoglobin level | 6 months

SECONDARY OUTCOMES:
the occurence of side effects (abdominal colics, constipation, or metallic taste) | 6 months
change in serum ferritin level | 6 months

OTHER OUTCOMES:
cost of treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Sayed, professor, Study Director — Cairo University
Locations (1):
- faculty of medicine, Cairo University, Cairo, Cairo Governorate, Egypt